CLINICAL TRIAL: NCT07298629
Title: Product Information Analysis and Clinical Verification - Clinical Verification of New Smart Health Medical Shoes/Insoles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202311043RIPA
Record Dates: First submitted 2025-11-21; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Pronated Foot
Keywords: 3D printed insoles; foot pressure; physical performance; motion analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D customized insole (Experimental)
  Interventions: Device: 3d printed insole

INTERVENTIONS:
Device: 3d printed insole — This study used 3D printer, producing customized insoles with selective laser sintering (SLS) technology.

SUMMARY:
As part of foot orthotics, insoles play a crucial role in adjusting biomechanical malalignments of the foot and regulating foot pressure. They are commonly used as a clinical tool for correcting foot problems. Currently, most customized insole manufacturing processes mainly depend on traditional or subtractive methods, highly dependent on the manual technology of the manufacturer, and the production capacity is constrained by working hours and cannot be manufactured in large quantities. Consequently, people often need to wait for one to two months with poor timeliness. The 3D printing insole fabrication process offers significant advantages in customization with high design flexibility and freedom. Utilizing microstructural zoning designs can better combine different regional characteristic requirements, thus closely addressing individual requirements. The purpose of this project is to validate the medical process after the initial development of the novel intelligent health medical insole and subsequently introduce the new intelligent health medical insole into clinical applications within medical institutions.

The project plans to recruit 30 participants with foot pain. Participants will be required to provide basic information and evaluated their foot condition. the Tiger Scan 3D full-foot scanning equipment will be used to capture the participants' 3D foot models. Insoles will be customized based on the assessment results, incorporating features such as heel cups, arch supports, and medial wedges. Relevant parameters will be uploaded to a RESTful API correction information platform. Then, the clinical recommendations for adjustment parameters will be output to a 3D printer, producing customized insoles with selective laser sintering (SLS) technology. The outcome assessments encompass short-term and long-term evaluations. Short-term assessments include kinematics and dynamic analysis, foot pressure distribution, physical performance, and foot morphology. Long-term assessments include pain levels, activities of daily living, and changes in quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Obvious medial arch collapse
2. Foot posture index (FPI) score of 6 or higher

Exclusion Criteria:

1. experience wearing custom-made insoles within the past 6 months;
2. experience of lower limb injury, surgery, acute infection, or other complications within the past 6 months
3. a body mass index (BMI) greater than 35;
4. rheumatoid arthritis;
5. cognitive impairment preventing obedience;
6. systemic diseases affecting the nervous, muscular, skeletal, or circulatory systems

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Foot pressure | Baseline, Week 1, Week 4
Foot functional Index | Baseline, Week 1, Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- School and Graduate Institute of Physical Therapy, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No